CLINICAL TRIAL: NCT04424121
Title: Cardiac CT, Calcium Scoring and ECG Stress Testing in Patients With Suspected Coronary Artery Disease: Precision Phenotyping and Financial Evaluation (The DATASET-PRECISE Randomized Trial)
Brief Title: CCTA, CACS and ECG Stress Testing in Patients With Suspected CAD: Precision Phenotyping and Financial Evaluation
Acronym: DATASET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Lefkos Stavros The Athens Clinic (Unknown); National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Georgios P Rampidis, MD, MSc, Academic Scholar, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DATASET PRECISE_01062020_03448
Record Dates: First submitted 2020-06-06; First posted 2020-06-09 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Stable Angina; Coronary Artery Disease; Atherosclerosis; Coronary Artery Calcification
Keywords: Coronary Computed Tomography Angiography; Coronary Artery Calcium Score; ECG Stress Test; Metabolomics; Precision Medicine; Artificial Intelligence; Machine Learning; Cost-Effectiveness Analysis; Clinical Decision Support Tool
MeSH Terms: conditions — Angina, Stable; Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Intervention Model Description: Open-label, 3-arm parallel randomized study
Masking Description: Open-label, 3-arm parallel randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of care plus ECG Stress Testing (No Intervention): Participants will be approached and randomized to receive standard care plus ECG-stress testing
- Standard of care plus ECG Stress Testing and CACS (No Intervention): Participants will be approached and randomized to receive standard care plus ECG-stress testing and coronary artery calcium scoring
- Standard of care plus CCTA (Active Comparator): Participants will be approached and randomized to receive standard care plus ≥ 64 multidetector coronary computed tomography angiography
  Interventions: Diagnostic Test: CCTA

INTERVENTIONS:
Diagnostic Test: CCTA — Coronary Computed Tomography Angiography
  Arms: Standard of care plus CCTA

SUMMARY:
The "DATASET-PRECISE", a 3-arm parallel randomized study, aims to provide new insights in risk stratification of patients with suspected CAD in the Greek population. The convergence of information derived from exercise ECG stress test, CACS, CCTA and metabolomic profiling in artificial intelligence algorithms describes in brief the main objective of this protocol. The design of the present proposal is based on current state-of-the-art literature, incorporating, however, additional innovative elements. It is about the first randomized study to be conducted in Greece, investigating the role of CCTA and CACS in CAD diagnosis and risk assessment. Moreover, the present protocol aims to integrate information on patients' metabolomic profiling. The process of the whole information by using artificial intelligence technology will lead to the development of new risk stratification algorithms, promoting further personalized diagnostic and therapeutic approach. Regarding Greece, this is the first prospectively enrolling medical database of this scale.

DETAILED DESCRIPTION:
Symptom-based pre-test probability (PTP) scores that estimate the likelihood of obstructive CAD in stable chest pain have moderate accuracy. Appreciating and integrating the myriad risk predictors in an individual patient is a challenge for the clinician. To date, efforts to improve risk-stratification by using CCTA have largely relied upon luminal stenosis severity. The emphasis placed on this variable over others is in alignment with prior studies using invasive coronary angiography but ignores an array of other parameters important in the CAD pathogenic process, including coronary artery geometry, coronary calcium content, plaque composition, and plaque burden. As an increasing number of CCTA variables along with all clinical and metabolomic variables affecting risk need to be considered, the complexity of assessment increases, making it more difficult for a clinician to draw an overall conclusion regarding risk in an individual patient. Furthermore, the potential influence of unexpected interactions between several weaker predictors in an individual patient is often overlooked. In this study, we are seeking to develop an Artificial Intelligence (AI)-based model, utilizing clinical and metabolomic risk factors, serum biomarkers, CCTA imaging biomarkers, coronary artery calcium score and ECG stress testing variables, to predict the presence and the complexity of CAD. Moreover, we are trying to introduce an easy to use, cost-effective, clinical decision supporting tool. In clinical practice, the utilization of such an approach could improve risk stratification and help guide downstream personalized management. Briefly, the research objectives of the study are: 1. predict the risk of obstructive coronary artery disease, 2. quantify the burden and complexity of coronary atherosclerosis, 3. evaluate the prognostic risk in individual patients with suspected CAD, 4. provide more accurate diagnosis and risk stratification, 5. provide an easy to use, cost-effective clinical decision support tool, 6. improve decisions in low to intermediate risk patients regarding the need for further testing such as cardiac SPECT and invasive coronary angiography, as well as for the need for preventive therapies and finally, compare three diagnostic strategies in patients with suspected CAD in terms of efficacy and cost-effectiveness.

The "DATASET-PRECISE" is a prospective, multi-center, open-label, 3-arm parallel randomized study. Following clinical consultation, participants will be approached and randomized 1:1:1 to receive standard care plus ECG-stress testing or standard care plus ECG-stress testing and CACS or standard care plus ≥ 64-multidetector CCTA and CACS (Collaborating Organizations: 1st Cardiology Department of AUTH, 1st Cardiology Department of NKUA, Lefkos Stavros-The Athens Clinic & Affidea Kozani Cardiac Imaging Center). Randomization will be conducted using a web-based system to ensure allocation concealment. The trial will enroll consecutive patients with stable symptoms and suspected CAD admitted to study clinical sites over a period of 12 months. Patients with a previous history of CAD and/or prior revascularization will be excluded. Subjects will undergo screening during the first day of examination, a 5ml blood sample will be collected one minute prior examination for metabolomic analysis (collaboration with the Lab. of Bioanalysis & Toxicology, School of Medicine, AUTH) and will be followed for 18 months afterwards. The overall recruitment period is expected to last 12 months. The estimated total duration of the study from first patient screened to last patient last visit is 30 months.

Based on previous studies for 80% power at a two-sided P value of 0.05, we will need to recruit about 250 patients per group to detect a relative reduction in the combined MACE rate (cardiac death, non-fatal myocardial infarction, revascularization or chest-pain rehospitalization) of 10% in the CCTA arm. A sample size of N = 900 patients is a pragmatic approach for such a first clinical study in the Greek population. Health service costs will be assigned to the type and intensity of resource use, measured by the number of diagnostic and therapeutic procedures or interventions, medications, hospital clinic attendances and hospitalization episodes from randomization to 18 months of follow-up. Costs will be attributed to the need for: 1. additional invasive or noninvasive imaging, 2. drug therapy, 3. coronary revascularization and 4. hospitalization for chest pain.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stable symptoms and low to intermediate probability of coronary artery disease (CAD) referred for evaluation
2. Patients without known history of CAD
3. Patients older than 18 years
4. Patients giving voluntary written consent to participate in the study
5. Subject is willing to comply with study follow-up requirements

Exclusion Criteria:

1. Patients with a previous history of CAD
2. Patients who refuse to give written consent for participation in the study
3. In the investigator's opinion, subject will not be able to comply with the follow-up requirements
4. Known pregnancy
5. Subject has a known allergy to contrast agent that cannot be adequately pre-medicated
6. Inability or unwilling to undergo computed tomography scanning, such as exceeding weight tolerance of scanner
7. Severe renal failure (estimated Glomerular Filtration Rate-eGFR <30 mL/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | 18 months
  Defined as cardiac death, non-fatal myocardial infarction or revascularization with percutaneous coronary intervention or coronary artery bypass graft surgery. Revascularization procedures within 6 weeks after the index CCTA will be excluded because they may be triggered by the CCTA findings per se
Chest-pain rehospitalization | 18 months
  Frequency (%) of chest-pain rehospitalization

SECONDARY OUTCOMES:
Frequency of angina [Seattle Angina Questionnaire (SAQ)] | 6 months
  The SAQ quantifies patients' physical limitations caused by angina, the frequency of and recent changes in their symptoms, their satisfaction with treatment, and the degree to which they perceive their disease to affect their quality of life. Scores range from 0 to 100, where higher scores indicate better function (less physical limitation, less angina and better quality of life)
Frequency of angina [Seattle Angina Questionnaire (SAQ)] | 12 months
  The SAQ quantifies patients' physical limitations caused by angina, the frequency of and recent changes in their symptoms, their satisfaction with treatment, and the degree to which they perceive their disease to affect their quality of life. Scores range from 0 to 100, where higher scores indicate better function (less physical limitation, less angina and better quality of life)
Frequency of angina [Seattle Angina Questionnaire (SAQ)] | 18 months
  The SAQ quantifies patients' physical limitations caused by angina, the frequency of and recent changes in their symptoms, their satisfaction with treatment, and the degree to which they perceive their disease to affect their quality of life. Scores range from 0 to 100, where higher scores indicate better function (less physical limitation, less angina and better quality of life)
Generic health status [Medical Outcomes Study 12-Item Short Form (SF-12)] | 12 months
  The Medical Outcomes Study 12-Item Short Form (SF-12) is a general health questionnaire and is computed using the scores of 12 questions ranging from 0 to 100, where 0 indicates the lowest level of health and 100 indicates the highest level of health

CONTACTS AND LOCATIONS:
Overall Officials: Haralambos Karvounis, Prof. in Cardiology, Study Chair — Aristotle University Of Thessaloniki; Georgios Giannakoulas, Prof. in Cardiology, Study Director — Aristotle University Of Thessaloniki; Periklis Kounatiadis, MD, PhD, Principal Investigator — Aristotle University Of Thessaloniki; Panagiotis Bamidis, Prof. in Bioinformatics, Principal Investigator — Aristotle University Of Thessaloniki; Georgios Rampidis, MD, MSc, Principal Investigator — Aristotle University Of Thessaloniki; Olga Deda, PhD, Principal Investigator — Aristotle University Of Thessaloniki; Antonios Billis, PhD, Principal Investigator — Aristotle University Of Thessaloniki
Locations (3):
- Greece (3):
  - Lefkos Stavros The Athens Clinic, Athens
  - National and Kapodistrian University of Athens, School of Medicine, Athens
  - Aristotle University of Thessaloniki, School of Medicine, Thessaloniki

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benz DC, Benetos G, Rampidis G, von Felten E, Bakula A, Sustar A, Kudura K, Messerli M, Fuchs TA, Gebhard C, Pazhenkottil AP, Kaufmann PA, Buechel RR. Validation of deep-learning image reconstruction for coronary computed tomography angiography: Impact on noise, image quality and diagnostic accuracy. J Cardiovasc Comput Tomogr. 2020 Sep-Oct;14(5):444-451. doi: 10.1016/j.jcct.2020.01.002. Epub 2020 Jan 13. PMID 31974008
- [Background] Benetos G, Buechel RR, Goncalves M, Benz DC, von Felten E, Rampidis GP, Clerc OF, Messerli M, Giannopoulos AA, Gebhard C, Fuchs TA, Pazhenkottil AP, Kaufmann PA, Grani C. Coronary artery volume index: a novel CCTA-derived predictor for cardiovascular events. Int J Cardiovasc Imaging. 2020 Apr;36(4):713-722. doi: 10.1007/s10554-019-01750-2. Epub 2020 Jan 1. PMID 31894527
- [Background] Rampidis GP, Benetos G, Benz DC, Giannopoulos AA, Buechel RR. A guide for Gensini Score calculation. Atherosclerosis. 2019 Aug;287:181-183. doi: 10.1016/j.atherosclerosis.2019.05.012. Epub 2019 May 10. No abstract available. PMID 31104809
- [Background] Knuuti J, Wijns W, Saraste A, Capodanno D, Barbato E, Funck-Brentano C, Prescott E, Storey RF, Deaton C, Cuisset T, Agewall S, Dickstein K, Edvardsen T, Escaned J, Gersh BJ, Svitil P, Gilard M, Hasdai D, Hatala R, Mahfoud F, Masip J, Muneretto C, Valgimigli M, Achenbach S, Bax JJ; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of chronic coronary syndromes. Eur Heart J. 2020 Jan 14;41(3):407-477. doi: 10.1093/eurheartj/ehz425. No abstract available. PMID 31504439
- [Background] Budoff MJ, Mayrhofer T, Ferencik M, Bittner D, Lee KL, Lu MT, Coles A, Jang J, Krishnam M, Douglas PS, Hoffmann U; PROMISE Investigators. Prognostic Value of Coronary Artery Calcium in the PROMISE Study (Prospective Multicenter Imaging Study for Evaluation of Chest Pain). Circulation. 2017 Nov 21;136(21):1993-2005. doi: 10.1161/CIRCULATIONAHA.117.030578. Epub 2017 Aug 28. PMID 28847895
- [Background] SCOT-HEART Investigators; Newby DE, Adamson PD, Berry C, Boon NA, Dweck MR, Flather M, Forbes J, Hunter A, Lewis S, MacLean S, Mills NL, Norrie J, Roditi G, Shah ASV, Timmis AD, van Beek EJR, Williams MC. Coronary CT Angiography and 5-Year Risk of Myocardial Infarction. N Engl J Med. 2018 Sep 6;379(10):924-933. doi: 10.1056/NEJMoa1805971. Epub 2018 Aug 25. PMID 30145934
- [Background] Hilvo M, Meikle PJ, Pedersen ER, Tell GS, Dhar I, Brenner H, Schottker B, Laaperi M, Kauhanen D, Koistinen KM, Jylha A, Huynh K, Mellett NA, Tonkin AM, Sullivan DR, Simes J, Nestel P, Koenig W, Rothenbacher D, Nygard O, Laaksonen R. Development and validation of a ceramide- and phospholipid-based cardiovascular risk estimation score for coronary artery disease patients. Eur Heart J. 2020 Jan 14;41(3):371-380. doi: 10.1093/eurheartj/ehz387. PMID 31209498
- [Background] von Felten E, Messerli M, Giannopoulos AA, Benz DC, Schwyzer M, Benetos G, Rampidis G, Patriki D, Kamani CH, Grani C, Fuchs TA, Pazhenkottil AP, Gebhard C, Kaufmann PA, Buechel RR. Potential of Radiation Dose Reduction by Optimizing Z-Axis Coverage in Coronary Computed Tomography Angiography on a Latest-Generation 256-Slice Scanner. J Comput Assist Tomogr. 2020 Mar/Apr;44(2):289-294. doi: 10.1097/RCT.0000000000000993. PMID 32195809